CLINICAL TRIAL: NCT05449210
Title: Reliability and Validity of Urdu Version of Parkinson's Disease Questionnaire in Pakistani Parkinson's Population
Brief Title: Urdu Version of Parkinson's Disease Questionnaire: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00237
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Quality of Life
Keywords: Parkinson's Disease Questionnaire-39; Parkinson's Disease; Reliability; Validity; Urdu Version
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the study , the researchers will investigate the reliability and validity of Urdu version Parkinson's Disease Questionnaire in Pakistani population having Parkinsonism

DETAILED DESCRIPTION:
The study is aimed to translate and culturally adapt Parkinson's Disease Questionnaire-39 into Urdu language and to investigate validity and reliability of Parkinson's Disease Questionnaire-39 in Parkinson's diseased patient among Pakistani population.The study will be a cross sectional survey in which non-probability purposive sampling technique will be used to enroll the participants into the study as per criteria.

The results of the study will help to establish an understanding of validity and reliability of Urdu version of Parkinson's Disease Questionnaire-39 with quality of life of Parkinson's Disease patients in Pakistani population having Parkinson's Disease. Reliability of the scale will be checked through internal consistency and test-retest methods. Cronbach's alpha value will be used to analyze internal consistency and for analyzing test-retest reliability an intraclass correlation coefficient with 195 patients will be used

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's Disease
2. Minimum age of 40 years
3. Minimum level of 5 years of education
4. A score equal to or greater than 23 on the Mini-Mental State Examination
5. Patient experiencing at least two of the three cardinal symptoms of idiopathic Pairkinson Disease (rigidity, resting tremor, and bradykinesia.)

Exclusion Criteria:

1. Patients with non-idiopathic Parkinsonian variants
2. Patients with a history of drug or alcohol abuse in the last two years
3. Patients with unstable medical problems that may place the patient at increased risk or may interfere with the assessment or treatment of Parkinson's
4. Neurological operation on the brain within one year prior to study entry

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson Disease in advanced age along tremors, rigidity and bradykinesia and postural abnormalities.will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Questionnaire | 12th Week
  The Parkinson's Disease Questionnaire checks the quality of life of patients suffering from Parkinson Disease

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No